CLINICAL TRIAL: NCT05738889
Title: Comparative Evaluation of Salivary Bisphenol-A Levels in Patients With Fixed Lingual, Hawley and Vacuum-formed Retainers
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, YAZGI AY UNUVAR, PhD, Assistant Professor, Aydin Adnan Menderes University
Other Study IDs: DHF-21010
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Orthodontic Retention
Keywords: Orthodontic retention; Bisphenol-A; lingual retainer; Hawley retainer; Vacuum formed retainer; essix plate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Patients with fixed lingual retainers applied with Bis-GMA containing composite: In the maxilla and mandible, the lingual surfaces of the anterior six teeth, including the canines, were roughened and bonded by applying 37.5% phosphoric acid for 30 seconds. Then, the retainer wire was adhered to the lingual surfaces of the teeth between the canine-canines in the maxilla and mandible, where a fixed lingual retainer will be applied, with a flowable composite adhesive containing Bis-GMA, with 10 seconds of illumination for 60 seconds for each tooth.
  Interventions: Device: Fixed lingual retainers applied with Bis-GMA containing composite
- Group 2: Patients with fixed lingual retainers applied with Bis-GMA-free composite: The lingual surfaces of the anterior six teeth, including the canines, in the maxilla and mandible were roughened by the application of 37.5% phosphoric acid for 30 seconds. Since the applied composite system is one-stage, no additional bond application was done. Fixed lingual retainer wire was applied with a Bis-GMA-free flowable composite adhesive with 60 seconds exposure for 10 seconds for each tooth.
  Interventions: Device: Fixed lingual retainers applied with Bis-GMA-free composite
- Group 3: Patients with vacuum-formed retainers: Impressions were taken with alginate impression material from the maxilla and mandible of the volunteers whose treatment was completed, and a model was obtained with a hard cast. On the models obtained, vacuum formed retainers were prepared with a vacuum forming machine. The use and care instructions of vacuum formed retainers were explained to the patient orally. vacuum formed retainers were used by the patient for 22 hours.
  Interventions: Device: Vacuum-formed retainers
- Group 4: Patients with hawley retainers: Impressions were taken with alginate impression material from the volunteers in the Hawley retainers group and a model was obtained with hard plaster. Wire elements were made on the model obtained and the appliance was prepared from transparent acrylic material. After the leveling and polishing processes were completed, the hawley retainers was attached to the mouth. It is stated that the appliance is used for 22 hours in 1 day. The use and care instructions of the Hawley retainers are explained to the patient.
  Interventions: Device: Hawley retainers

INTERVENTIONS:
Device: Fixed lingual retainers applied with Bis-GMA containing composite — Bonding materials of fixed lingual retainers applied with Bis-GMA containing composite
  Other Names: Reliance Orthodontic Gel Etching Agent, Illinois, USA; American Orthodontics Brace Paste MTP primer, Wisconsin, USA; Reliance Orthodontic Bond-A-Braid, Illinois, USA; Reliance Orthodontic Flow Tain Low Viscosity W/TIPS, Illinois, USA
  Groups: Group 1: Patients with fixed lingual retainers applied with Bis-GMA containing composite
Device: Fixed lingual retainers applied with Bis-GMA-free composite — Bonding materials of fixed lingual retainers applied with Bis-GMA-free composite
  Other Names: Reliance Orthodontic Gel Etching Agent, Illinois, USA; Reliance Orthodontic Bond-A-Braid, Illinois, USA; GC Ortho Connect Flow, Tokyo, Japan
  Groups: Group 2: Patients with fixed lingual retainers applied with Bis-GMA-free composite
Device: Vacuum-formed retainers — vacuum-forming machine and vacuum formed plates
  Other Names: Supplies Atmos Thermoforming Material 0.40 inç, USA; Dentsply Sirona, USA
  Groups: Group 3: Patients with vacuum-formed retainers
Device: Hawley retainers — Acrylic based hawley retainers
  Other Names: Dentaurum Orthocryl, Ispringen, Germany
  Groups: Group 4: Patients with hawley retainers

SUMMARY:
The aim of this study; to measure the BPA release amount of fixed lingual retainers applied with Bis-GMA-containing composite , fixed lingual retainers applied with Bis-GMA-free composite, vacuum-formed and hawley retainers which used for retention after orthodontic treatment to evaluate whether they are risk factors for the patient and to compare BPA releases.

Study method and data collection techniques: In this study, individuals will be selected from the patients who will be treated at Aydın Adnan Menderes University Faculty of Dentistry, Department of Orthodontics between July 2021 and July 2022, whose orthodontic treatment will be completed. These patients will be randomly divided into four groups according to the type of retention appliance to be chosen: those who are applied a fixed lingual retainer with a bis-GMA-containing composite, those with a fixed lingual retainer with a bis-GMA-free composite, those with an vacuum formed retainers, and those with a hawley retainers. After the debonding of the fixed attachments at the end of the treatment appointment, the retention appliances will be applied 1 day later so that BPA, which is released from the resin adhesives used to bond the attachments, does not affect the study data. Saliva samples will be taken from the patients before the appliance is inserted, 1 hour, 7 days and 30 days after the appliance is inserted.

DETAILED DESCRIPTION:
Patients who are scheduled to complete their orthodontic treatment between July 2021 and July 2022 and will be debonded will be included in the study. Inclusion criteria for the study; not to have any systemic diseases, not to smoke, not to work in jobs where they will be exposed to chronic BPA release, such as gas station-construction site or acrylic-related jobs. Selected patients will be randomly divided into four groups. Randomization will be done through the website www.random.org. Fixed lingual retainer applied with composite containing Bis-GMA will be applied in the first group, fixed lingual retainer applied with composite without Bis-GMA in the second group, vacuum formed retainers in the third group and hawley retainers in the fourth group. 120 patients, including 30 individuals in each group, will be included in the study. The number of men and women in each group will be equal. Patients who have undergone debonding will be given an appointment to wear retention appliances one day later. Patients will be advised to brush their teeth routinely, including the appointment day, and not to consume any food or drink at least 2 hours before the application. In addition, due to the effect of many drugs on salivary secretion, if patients use drugs, they will be told to take them at least 8 hours before the application. Saliva samples for BPA release will be taken before appliance insertion, 1 hour after, 7 days and 30 days after insertion. Samples taken will be stored in polypropylene tubes. All samples taken will be stored at -80 degrees until analysis. The sample will be processed by mixing 5ml saliva with an equal amount of ethanol and vortexing it. It will be centrifuged at 3000 rpm for 15 minutes. The ultimately processed sample will be injected into the instrument and analyzed by liquid chromatography.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages 10-18
* absence of any systemic disease
* good oral hygiene
* completion of orthodontic treatment
* non smoker
* Not working in jobs where they will be exposed to chronic BPA release, such as gas station construction site or acrylic related jobs

Exclusion Criteria:

* be under 10 years or over 18 years
* any systemic disease
* poor oral hygiene
* ıncomplete orthodontic treatment
* being a smoker
* working in jobs where they will e exposed to chronic BPA release, such as gas station construction site or acrylic related jobs

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Men and women patients aged between 10-18 years who have completed orthodontic treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
Bisphenol-A amount in saliva before applying a retainer with bis-GMA-containing composite | 1 day after debonding and before retention appliance to 1 month.
  The main purpose of this thesis study is to determine the appliance with the least BPA release by comparing the Bisphenol-A(BPA) release levels from lingual retainers, vacuum formed retainers and hawley retainers used for retention after orthodontic treatment. Saliva samples were taken from volunteers at regular intervals, a total of 4 times. First example; One day after debonding, before applying the retention appliance, the second sample; One hour after the retention appliance was applied, the third sample was taken 1 week later and the fourth sample 1 month later. Analysis of the change in BPA was done.
Bisphenol-A amount in saliva before applying a retainer with bis-GMA-free composite | 1 day after debonding and before retention appliance to 1 month.
  The main purpose of this thesis study is to determine the appliance with the least BPA release by comparing the Bisphenol-A(BPA) release levels from lingual retainers, vacuum formed retainers and hawley retainers used for retention after orthodontic treatment. Saliva samples were taken from volunteers at regular intervals, a total of 4 times. First example; One day after debonding, before applying the retention appliance, the second sample; One hour after the retention appliance was applied, the third sample was taken 1 week later and the fourth sample 1 month later. Analysis of the change in BPA was done.
Bisphenol-A amount in saliva before applying vacuum formed retainer | 1 day after debonding and before retention appliance to 1 month.
  The main purpose of this thesis study is to determine the appliance with the least BPA release by comparing the Bisphenol-A(BPA) release levels from lingual retainers, vacuum formed retainers and hawley retainers used for retention after orthodontic treatment. Saliva samples were taken from volunteers at regular intervals, a total of 4 times. First example; One day after debonding, before applying the retention appliance, the second sample; One hour after the retention appliance was applied, the third sample was taken 1 week later and the fourth sample 1 month later. Analysis of the change in BPA was done.
Bisphenol-A amount in saliva before applying hawley retainer | 1 day after debonding and before retention appliance to 1 month.
  The main purpose of this thesis study is to determine the appliance with the least BPA release by comparing the Bisphenol-A(BPA) release levels from lingual retainers, vacuum formed retainers and hawley retainers used for retention after orthodontic treatment. Saliva samples were taken from volunteers at regular intervals, a total of 4 times. First example; One day after debonding, before applying the retention appliance, the second sample; One hour after the retention appliance was applied, the third sample was taken 1 week later and the fourth sample 1 month later. Analysis of the change in BPA was done.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University Faculty of Dentistry, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Raghavan AS, Pottipalli Sathyanarayana H, Kailasam V, Padmanabhan S. Comparative evaluation of salivary bisphenol A levels in patients wearing vacuum-formed and Hawley retainers: An in-vivo study. Am J Orthod Dentofacial Orthop. 2017 Mar;151(3):471-476. doi: 10.1016/j.ajodo.2016.07.022. PMID 28257731
- [Result] Manoj MK, Ramakrishnan R, Babjee S, Nasim R. High-performance liquid chromatography analysis of salivary bisphenol A levels from light-cured and chemically cured orthodontic adhesives. Am J Orthod Dentofacial Orthop. 2018 Dec;154(6):803-808. doi: 10.1016/j.ajodo.2018.02.008. PMID 30477778
- [Result] Eliades T, Voutsa D, Sifakakis I, Makou M, Katsaros C. Release of bisphenol-A from a light-cured adhesive bonded to lingual fixed retainers. Am J Orthod Dentofacial Orthop. 2011 Feb;139(2):192-5. doi: 10.1016/j.ajodo.2009.12.026. PMID 21300247
- [Result] Sasaki N, Okuda K, Kato T, Kakishima H, Okuma H, Abe K, Tachino H, Tuchida K, Kubono K. Salivary bisphenol-A levels detected by ELISA after restoration with composite resin. J Mater Sci Mater Med. 2005 Apr;16(4):297-300. doi: 10.1007/s10856-005-0627-8. PMID 15803273
- [Result] Kang YG, Kim JY, Kim J, Won PJ, Nam JH. Release of bisphenol A from resin composite used to bond orthodontic lingual retainers. Am J Orthod Dentofacial Orthop. 2011 Dec;140(6):779-89. doi: 10.1016/j.ajodo.2011.04.022. PMID 22133942
- [Result] Eliades T, Hiskia A, Eliades G, Athanasiou AE. Assessment of bisphenol-A release from orthodontic adhesives. Am J Orthod Dentofacial Orthop. 2007 Jan;131(1):72-5. doi: 10.1016/j.ajodo.2006.08.013. PMID 17208109